CLINICAL TRIAL: NCT02068391
Title: Achieving Brain Benefits in Covert Stroke Through Aerobic Exercise
Brief Title: Recovery Improved in Covert Stroke With Exercise
Acronym: RISE-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Toronto Rehabilitation Institute (Other)
Responsible Party: Principal Investigator, Dr. Bradley MacIntosh, Imaging Scientist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: RISE2-2014-312185
Record Dates: First submitted 2014-02-19; First posted 2014-02-21 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Cerebral Small Vessel Diseases
Keywords: covert stroke; cerebral blood flow; grey matter; attention; executive function; aerobic exercise
MeSH Terms: conditions — Cerebral Small Vessel Diseases | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): This group will perform the 'Exercise Program' for months 0 to 6, and will be unsupervised for months 7 to 12.
  Interventions: Behavioral: Exercise Program
- Stretching (Active Comparator): This group will perform the 'Stretching Program' for months 0 to 6, and the 'Exercise Program' for months 7 to 12.
  Interventions: Behavioral: Stretching Program; Behavioral: Exercise Program

INTERVENTIONS:
Behavioral: Stretching Program — The 'Stretching Program' will teach stretching for the upper and lower limbs, and the trunk, as well as breathing exercises for relaxation. Supervised group activities will be performed once per week (45 minutes) and self-directed stretching will be encouraged 4 days per week and monitored by an activity journal. The intensity of stretching and number of stretches will be progressed every 2 weeks. Heart rate and perceived exertion will be monitored. The program will last 6 months.
  Arms: Stretching
Behavioral: Exercise Program — The 'Exercise Program' will prescribe specific aerobic exercise to the participants. Supervised group exercise will be performed once per week (60 minutes) and self-directed exercise will be encouraged 4 days per week and monitored by an activity journal. The initial walking prescription will be set at ~1.6 km and an intensity equivalent to the anaerobic threshold and/or 60% of peak oxygen uptake. Progressions will be made every 2 weeks, increasing distance to a maximum of 6.4 km and then increasing to a max intensity of 80% of peak oxygen uptake and/or max duration of 60 minutes. Heart rate and perceived exertion will be monitored. The program will last 6 months.

SUMMARY:
Silent ischemic, also known as "covert stroke vascular disease" (CSVD), contributes to neurological deficits that are caused by damage to small blood vessels in the brain. CSVD occurs six to ten times more often that an acute stroke. It is misleading to think, however, that CSVD is an inevitable part of "getting old" because people with CSVD are at high risk of developing an acute stroke or dementia. In fact, people with more CSVD lesion volume are more likely to develop day to day problems in planning, decision-making and speed of thinking. Unfortunately, there are no proven therapies designed to address CSVD. We propose to test whether aerobic exercise is an intervention that can combat CSVD because the disease is fundamentally a blood flow problem that may be improved by aerobic exercise. We will recruit CSVD adults with moderate to severe lesion burden and use magnetic resonance imaging (MRI) to study the brain in terms of structure, perfusion and function. Participants will be randomly assigned to either our established aerobic exercise program or a control stretching program. Both groups will take part in lab exercise sessions, which are designed to monitor progress and assess adherence to the program. The duration and intensity of their exercise will increase as participants progress. We will use activity log books, phone calls and extra "booster" exercise sessions, as needed, to maximize retention and adherence. We aim to show that aerobic exercise increases cerebral blood flow (CBF) in frontal-subcortical grey matter, supports regional tissue growth, and improves cognitive function in CSVD adults with substantial risk of acute stroke and dementia. A positive outcome of this research will provide strong support for additional clinical trials aimed at sustaining cognition and maintaining independent living.

ELIGIBILITY:
Inclusion Criteria:

* Covert stroke: white matter hyperintensities of presumed vascular origin
* Ability to walk for 10 minutes without assistance from another person
* Fluent in English
* Ability to consent

Exclusion Criteria:

* Highly fit individuals exercising ≥ 150 minutes per week
* Dementia
* Multiple Sclerosis
* Disabling stroke (ischemic or hemorrhagic)
* Major concurrent illness (e.g. chronic obstructive lung disorder, current or metastatic cancer, chronic kidney disease)
* Major psychiatric illness (e.g. bipolar, schizophrenia, major depression)
* Contraindications to MRI scanning (e.g. claustrophobia, implants, prostheses, metallic fragments)
* Contraindications to exercise (participants must have medical clearance to exercise from their attending physician)
* Recent change in health status (e.g. hospitalization within past month)

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2018-03-07 (Actual); Study Completion 2018-09-12 (Actual)

PRIMARY OUTCOMES:
Change in cerebral blood flow from baseline to 6 months | 6 months
  Pseudo-continuous arterial spin labeling MRI
Change in brain structure from baseline to 6 months | 6 months
  Cortical and subcortical grey matter density using structural MRI

SECONDARY OUTCOMES:
Change in brain activity related to attention and executive control tasks from baseline to 6 months | 6 months
  Blood oxygenation level dependent MRI

OTHER OUTCOMES:
Change in white matter integrity from baseline to 6 months | 6 months
  Diffusion tensor imaging (DTI) MRI
Change in aerobic fitness from baseline to 6 months | 6 months
  Peak oxygen uptake
Change in aerobic fitness from 6 to 12 months | 12 months
  Peak oxygen uptake
Change in autonomic function from baseline to 6 months | 6 months
  Heart rate variability
Change in autonomic function from 6 to 12 months | 12 months
  Heart rate variability
Change in arterial stiffness from baseline to 6 months | 6 months
  Carotid-femoral pulse wave velocity
Change in arterial stiffness from 6 to 12 months | 12 months
  Carotid-femoral pulse wave velocity
Change in executive function from baseline to 6 months | 6 months
  Trail Making Test
Change in executive function from 6 to 12 months | 12 months
  Trail Making Test
Change in balance from baseline to 6 months | 6 months
  Spatial-temporal synchronization of center of pressure
Change in balance from 6 to 12 months | 12 months
  Spatial-temporal synchronization of center of pressure
Change in dual task gait from baseline to 6 months | 6 months
  Comparison of normal gait to gait with verbal math challenge
Change in dual task gait from 6 to 12 months | 12 months
  Comparison of normal gait to gait with verbal math challenge
Change in grip strength from baseline to 6 months | 6 months
  Maximum grip strength with dynamometer
Change in grip strength from 6 to 12 months | 12 months
  Maximum grip strength with dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Bradley MacIntosh, PhD, Principal Investigator — Sunnybrook Research Institute
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided